CLINICAL TRIAL: NCT04102566
Title: Optimizing Pain Control in Transurethral Resection of the Prostate
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Benaroya Research Institute (Other)
Collaborators: Virginia Mason Hospital/Medical Center (Other)
Responsible Party: Principal Investigator, Una Lee, Principal Investigator and Attending urologist, Benaroya Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB17-098
Record Dates: First submitted 2019-09-23; First posted 2019-09-25 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Pain; BPH With Urinary Obstruction; BPH With Urinary Obstruction With Other Lower Urinary Tract Symptoms
Keywords: postoperative pain; Transurethral resection of the prostate; Multimodal pain control
MeSH Terms: conditions — Pain; Pain, Postoperative | interventions — Ibuprofen; Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of care arm (No Intervention): The standard of care group will group will receive the following regimen while inpatient:
  * 2% topical lidocaine gel applied to catheter tip as needed for pain, maximum dose of 600mg in 12 hours
  * Acetaminophen 1000mg every 8 hours standing
  * Oxycodone 5mg PO every 4 hours as needed pain
  * Phenazopyridine 100mg TID as needed for urinary burning
  * Senna 1 tab every 12 hours
  * Miralax 17g powder once daily as needed for constipation
  The standard of care group will get the following prescriptions on discharge:
  * Oxycodone 5mg every 4 hours as needed pain - 15 tabs
  * Acetaminophen 1000mg every 8 hours standing for two days then as needed
  * Phenazopyridine 100mg TID as needed for urinary burning - 9 tabs
  * Senna 1 tab every 12 hours - 10 tabs
- Multi-modal group (Experimental): The multi-modal group will receive the following regimen while inpatient:
  * 2% topical lidocaine gel applied to catheter tip as needed for pain, maximum dose of 600mg in 12 hours
  * Acetaminophen 1000mg every 8 hours standing
  * Ibuprofen 600mg every 6 hours standing
  * Oxycodone 5mg PO every 4 hours as needed pain
  * Phenazopyridine 100mg TID as needed for urinary burning
  * Senna 1 tab every 12 hours
  * Miralax 17g powder once daily as needed for constipation
  * Patient Education (Figures 2 & 3)
  The multi-modal group will receive the following prescriptions on discharge:
  * Acetaminophen 1000mg every 8 hours standing for two days then as needed - 30 tabs
  * Ibuprofen 600mg every 8 hours standing for two days then as needed - 30 tabs
  * Phenazopyridine 100mg TID as needed for urinary burning - 9 tabs
  * Senna 1 tab every 12 hours - 10 tabs
  Interventions: Drug: Ibuprofen 600 mg; Behavioral: Education

INTERVENTIONS:
Drug: Ibuprofen 600 mg — We'll be adding ibuprofen while trying to limit oxycodone use while hospitalized. Patients will not be discharged with a narcotic.
  Arms: Multi-modal group
Behavioral: Education — We'll be adding education to patient's post-operative instructions to aid in their pain control management.
  Arms: Multi-modal group

SUMMARY:
The purpose of this study is to develop a multi-modal protocol for pain management after TURP that minimizes opioid use. The investigators hypothesize this approach will provide non-inferior pain control to the current standard of care which includes opioids as the primary agent. The investigators believe this is an important step in reducing the opioid epidemic in surgical patients.

DETAILED DESCRIPTION:
In our study, the investigators will randomize TURP patients to standard of care versus a multi-modal protocol. Multi-modal pain control is defined as: "analgesia that combines 2 or more agents that act by different mechanisms to provide analgesia with better pain relief and less opioids". In addition, patients in the intervention arm will receive education regarding pain control and opioid use. The investigators aim to demonstrate non-inferior pain control with this approach. The investigators hope this will inform new guidelines for pain control after TURP, minimize opioid use in this patient population, and educate physicians and patients on providing excellent pain control while minimizing the risks of opioid use. The investigators believe this could ultimately serve as a model for other endoscopic urologic procedures as well.

ELIGIBILITY:
Inclusion Criteria:

* Are identified as candidates for TURP
* Are 18 years of age or greater
* Are proficient in English

Exclusion Criteria:

* Have filled an opioid prescription in the last 2 months
* Have an allergy to a medication included in the protocol
* Have a history of pelvic radiation
* Have renal failure (Serum Cr > 2.0 mg/dl), peptic ulcer disease, history of gastric bypass, cirrhosis, or other contraindication precluding use of NSAID's
* Have liver failure, hepatitis, or alcohol abuse which precludes use of acetaminophen

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-12-08 (Actual); Primary Completion 2019-10-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Opioid Consumption | PACU-72 hours
  Total opioid utilization
Pain Scores | PACU-72 hours
  Numerical Rating Scale Pain Scores (Range: 0-10, where 0 is no pain and 10 is the worst pain)

SECONDARY OUTCOMES:
Presence of a foley catheter at discharge. | 0-48hours
  Was the patient discharged with a Foley catheter?
Presence of narcotic side effects | 48 hours after discharge
  nausea/vomiting, pruritus, constipation, dizziness or feelings of sedation
Were there any post-operative complications | 0-48 hours
  Any complications post-operatively that occurred in the immediate post-operative setting.

CONTACTS AND LOCATIONS:
Locations (1):
- Virginia Mason Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers. IPD will be used solely for this study cohort and protocol.

REFERENCES:
- [Background] Alam A, Gomes T, Zheng H, Mamdani MM, Juurlink DN, Bell CM. Long-term analgesic use after low-risk surgery: a retrospective cohort study. Arch Intern Med. 2012 Mar 12;172(5):425-30. doi: 10.1001/archinternmed.2011.1827. PMID 22412106
- [Background] Sun EC, Darnall BD, Baker LC, Mackey S. Incidence of and Risk Factors for Chronic Opioid Use Among Opioid-Naive Patients in the Postoperative Period. JAMA Intern Med. 2016 Sep 1;176(9):1286-93. doi: 10.1001/jamainternmed.2016.3298. PMID 27400458
- [Background] Hill MV, Stucke RS, McMahon ML, Beeman JL, Barth RJ Jr. An Educational Intervention Decreases Opioid Prescribing After General Surgical Operations. Ann Surg. 2018 Mar;267(3):468-472. doi: 10.1097/SLA.0000000000002198. PMID 28267689
- [Background] Hill MV, McMahon ML, Stucke RS, Barth RJ Jr. Wide Variation and Excessive Dosage of Opioid Prescriptions for Common General Surgical Procedures. Ann Surg. 2017 Apr;265(4):709-714. doi: 10.1097/SLA.0000000000001993. PMID 27631771
- [Background] Kose O, Saglam HS, Altun ME, Sonbahar T, Kumsar S, Adsan O. Prilocaine irrigation for pain relief after transurethral resection of the prostate. J Endourol. 2013 Jul;27(7):892-5. doi: 10.1089/end.2013.0001. Epub 2013 Jun 12. PMID 23565930
- [Background] American Society of Anesthesiologists Task Force on Acute Pain Management. Practice guidelines for acute pain management in the perioperative setting: an updated report by the American Society of Anesthesiologists Task Force on Acute Pain Management. Anesthesiology. 2012 Feb;116(2):248-73. doi: 10.1097/ALN.0b013e31823c1030. No abstract available. PMID 22227789
- [Background] Dowell D, Haegerich TM, Chou R. CDC Guideline for Prescribing Opioids for Chronic Pain--United States, 2016. JAMA. 2016 Apr 19;315(15):1624-45. doi: 10.1001/jama.2016.1464. PMID 26977696
- [Background] Maughan BC, Hersh EV, Shofer FS, Wanner KJ, Archer E, Carrasco LR, Rhodes KV. Unused opioid analgesics and drug disposal following outpatient dental surgery: A randomized controlled trial. Drug Alcohol Depend. 2016 Nov 1;168:328-334. doi: 10.1016/j.drugalcdep.2016.08.016. Epub 2016 Sep 20. PMID 27663358